CLINICAL TRIAL: NCT06756048
Title: Study of the Effects of Rhomboid Intercostal Block on Acute Postoperative Pain Management and Chronic Pain Incidence in Patients Undergoing Oncologic Breast Surgery
Brief Title: Effects of Rhomboid Intercostal Block on Postoperative Pain Management and Chronic Pain Incidence in Mastectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Kamil Darcin, Assoc. Prof., Koç University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023.391.IRB1.138
Record Dates: First submitted 2024-11-26; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Mastectomy; Rhomboid Intercostal Block; Chronic Pain Following Surgical Procedure for Cancer
Keywords: mastectomy; rhomboid intercostal block; chronic pain; chronic pain following surgical procedure for cancer; regional anesthesia; bupivacaine
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Group RIB: patients in this group will receive rhomboid intercostal block prior to mastectomy (any breast surgery due to a mass) Group Control: patients in this group will not receive any methods of regional anesthesia prior to mastectomy (any breast surgery due to a mass)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allocated to Intervention (Rhomboid Intercostal Block) (Experimental): Group I: RIB In the first group (Group RIB), patients will receive a Rhomboid Intercostal Block immediately before the induction of general anesthesia. The procedure will be performed with the patient sitting upright and premedicated with anxiolytics. Using ultrasound guidance, a 50 mm block needle will be inserted into the auscultatory triangle (interfascial plane located lateral to the erector spinae muscle, beneath the rhomboid major, and over the intercostal nerves). A total of 20 ml of 0.25% bupivacaine will be administered at this site.
  If the surgery is unilateral, the RIB will be applied only on the surgical side. For bilateral surgeries, 20 ml of bupivacaine will be administered to each side.
  Interventions: Procedure: Rhomboid Intercostal Nerve Block
- Allocated to No Intervention (Control Group) (No Intervention): Group II: Control Group In the second group (Control Group), patients will undergo the surgical procedure without receiving a Rhomboid Intercostal Block (RIB) or any other regional anesthesia technique. Standard general anesthesia protocols will be followed for these patients, and postoperative pain management will be conducted using systemic analgesics according to the institution's routine practice.

INTERVENTIONS:
Procedure: Rhomboid Intercostal Nerve Block — Following standard ASA monitoring, patients were positioned on the surgical table with their backs facing the operator. Skin antisepsis was achieved using povidone. A high-frequency 8-18 MHz linear ultrasound probe was used.
  After palpating the rhomboid muscles and intercostal spaces at the T6-T7 levels, the medial border of the scapula and the vertebral column were identified. The ultrasound probe was placed horizontally along the medial border of the scapula. Using ultrasound guidance, the ribs, rhomboid muscles, intercostal muscles, and pleura were visualized. Once these anatomical structures were clearly identified, a 50 mm, 22G regional block needle was advanced in-plane from caudal to cranial under ultrasound guidance until the interfascial plane beneath the rhomboid muscles was reached and total of 20 ml of 0.25% bupivacaine (Marcaine® 0.5%, AstraZeneca PLC, London, UK) was injected.
  Arms: Allocated to Intervention (Rhomboid Intercostal Block)

SUMMARY:
The goal of this clinical trial is to evaluate the effects of the Rhomboid Intercostal Block (RIB) on postoperative chronic pain prevalence at 3 months (primary outcome) and on acute pain control, total opioid consumption, and the incidence of opioid-related side effects within the first 24 hours (secondary outcomes) in patients undergoing elective mastectomy surgery.

The main questions it aims to answer are:

Does the application of RIB reduce the prevalence of chronic pain at 3 months postoperatively? Does RIB improve acute pain control and reduce opioid consumption and related side effects in the first 24 hours postoperatively? Researchers will compare patients who receive RIB under general anesthesia to those who do not receive the block to determine its effectiveness in reducing chronic pain prevalence, acute pain scores, and opioid-related outcomes.

DETAILED DESCRIPTION:
Primary Outcome Measures

The primary outcome is the prevalence of chronic pain at 3 months in patients undergoing mastectomy surgery. For patients reporting pain, additional parameters will be assessed, including:

Pain characteristics: location, frequency, intensity, and radiation. Factors that exacerbate or alleviate pain. Impact of pain on quality of life (measured on a 1-5 scale). Types and quantities of analgesics used. Secondary Outcome Measures

Acute Pain Scores:

Pain levels at 1, 6, 12, and 24 hours postoperatively at rest, measured using the Numeric Rating Scale (NRS).

Opioid Consumption and Side Effects:

Total opioid consumption (morphine and tramadol) within the first 24 hours postoperatively.

Incidence of opioid-related side effects, such as nausea, vomiting, and pruritus.

Patient Satisfaction and Sleep Quality:

Satisfaction with the analgesic method (e.g., very satisfied, satisfied, neutral, dissatisfied, very dissatisfied).

Sleep quality ratings (very good, good, moderate, poor, very poor). Willingness to use the same analgesic method again (yes/no).

Chronic Pain Impact on Daily Life (for patients with pain at 3 months):

Degree of limitation in physical activities, household/work tasks, and social life (scored on a scale from 0 = no limitation to 5 = constant limitation).

Impact on psychological well-being (scored on a scale from 0 = no impact to 5 = constant impact).

Study Design and Participants This prospective, randomized, controlled study will be conducted at Koç University Hospital. Participants will include 90 patients undergoing elective mastectomy surgery, aged 18-80 years, and classified as ASA I-III according to the American Society of Anesthesiologists. Written informed consent will be obtained from all participants.

The sample size calculation was based on a 2020 meta-analysis reporting a 59% prevalence of chronic pain at 3 months in patients without any regional block. Using select-statistics.co.uk software, with a two-proportion sample test, a 50% reduction in chronic pain prevalence was considered significant. With a p-value of 0.05 and 80% power, 43 patients per group were required. To increase robustness and account for potential dropouts, 45 patients per group (90 total) will be enrolled.

Randomization and Blinding: Participants will be randomized into two groups using randomizer.org software. RIB will be performed before induction of general anesthesia. No blinding will be performed due to the nature of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing one of the following procedures: benign mass excisions, modified radical mastectomies (MRM), simple total mastectomies, nipple-sparing mastectomies, or skin-sparing mastectomies, regardless of additional procedures such as sentinel lymph node biopsy (SLNB), axillary lymph node dissection (ALND), or implant placement.

Exclusion Criteria:

* Patients undergoing breast augmentation, reduction, or mammoplasty without a mass.
* Patients with a BMI > 35.
* Emergency cases.
* Patients with bleeding diathesis.
* Known allergy to medications used in the study.
* Patients with asthma.
* Patients diagnosed with chronic kidney failure.
* Pregnant or lactating patients.
* Patients with chronic opioid use.
* Patients with cooperation issues or inadequate communication ability.
* Male patients.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 90 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Chronic pain incidence at postoperative third month | from enrollment (surgery day) to the end of postoperative third month.
  participants will receive a phone call from the researcher at the end of third postoperative period. They will be asked 'are you experiencing any remaining pain' and their responses will be recorded as yes or no. Patients who respond yes will be calculated between groups to find the incidence of chronic pain.

SECONDARY OUTCOMES:
total morphine consumption at postoperative 24 hours | from enrollment to end of first postoperative day
  patients will be given a patient controlled analgesia device with no infusion, 1 mg morphine bolus and 10 minutes lock time. At 24.hour visit, their total morphine consumption will be recorded and analyzed in between groups for any statistical difference.
Postoperative pain levels with Numeric Rating Scale on 1st, 6th, 12th and 24th hours | from enrollment to end of first postoperative day
  Participants NRS pain scores at rest will be recorded for postoperative 1., 6., 12. and 24. hours at visits.
  They will be asked "on a scale of 0 (no pain) to 10 (worst pain imaginable), how would you rate your level of pain now?" and their answers will be recorded.
  Numeric Rating Scale is a scale from 0 to 10, 0-1-2-3-4-5-6-7-8-9-10 has 11 possible answers and higher numbers mean worse pain.
Postoperative nausea and vomiting incidence | from enrollment to end of first postoperative day
  patients will be monitorized for any opioid related side effects, mainly nausea and vomiting. If any respiratory depression, pruritus occurs it will also be recorded. groups will be compared for opioid related side effect incidence (nausea and vomiting)
Limitation on Daily Activities | from enrollment (surgery day) to the end of postoperative third month.
  At 3 months postoperatively, for patients experiencing pain, secondary outcome measures will include the degree of limitation in physical activities. Patients will be asked "how much your pain limits your daily activities" and will be asked to rate it from 0 to 5.
  0 (no limitation)
  1. (rarely limits)
  2. (sometimes limits)
  3. (usually limits)
  4. (mostly limits)
  5. (constant limitation). Social Life: Assessed on a scale from 0 (no limitation) to 5 (constant limitation).
  Psychological Well-Being: Impact on psychological well-being will be evaluated on a scale from 0 (no impact) to 5 (constant impact).
  These measures aim to evaluate the broader effects of pain on patients' quality of life and functional outcomes.
Household/Work Activities | from enrollment (surgery day) to the end of postoperative third month.
  At 3 months postoperatively, for patients experiencing pain, secondary outcome measures will include the degree of limitation in physical activities. Patients will be asked "how much your pain limits your household or work activities" and will be asked to rate it from 0 to 5.
  0 (no limitation)
  1. (rarely limits)
  2. (sometimes limits)
  3. (usually limits)
  4. (mostly limits)
  5. (constant limitation). These measures aim to evaluate the broader effects of pain on patients' quality of life and functional outcomes.
Social Life | from enrollment (surgery day) to the end of postoperative third month.
  At 3 months postoperatively, for patients experiencing pain, secondary outcome measures will include the degree of limitation in social life. Patients will be asked "how much your pain limits your social life" and will be asked to rate it from 0 to 5.
  0 (no limitation)
  1. (rarely limits)
  2. (sometimes limits)
  3. (usually limits)
  4. (mostly limits)
  5. (constant limitation). These measures aim to evaluate the broader effects of pain on patients' quality of life and functional outcomes.
Psychological Well Being | from enrollment (surgery day) to the end of postoperative third month.
  At 3 months postoperatively, for patients experiencing pain, secondary outcome measures will include the degree of limitation in social life. Patients will be asked "how much your pain limits your psychological well being" and will be asked to rate it from 0 to 5.
  0 (no limitation)
  1. (rarely limits)
  2. (sometimes limits)
  3. (usually limits)
  4. (mostly limits)
  5. (constant limitation). These measures aim to evaluate the broader effects of pain on patients' quality of life and functional outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Gürkan, Prof., Study Director — Koc University Medical School
Locations (1):
- Koc University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected through the trial can be shared with third parties upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: The IPD and supporting information will be available to share at the end of enrollment period and upon completion of third month pain data (27 November 2024). The information will be available for two years (until 27 November 2026)
Access Criteria: The IPD can be received from Dr. Belitsu Salgın (assistant investigator) and Assoc. Prof. Dr. Kamil Darçın (Investigator) upon reasonable request (for a medical research and improvement purpose). all data and statistical test data is available at our records.

REFERENCES:
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Harkouk H, Fletcher D, Martinez V. Paravertebral block for the prevention of chronic postsurgical pain after breast cancer surgery. Reg Anesth Pain Med. 2021 Mar;46(3):251-257. doi: 10.1136/rapm-2020-102040. Epub 2021 Jan 7. PMID 33414157
- [Background] Wang L, Cohen JC, Devasenapathy N, Hong BY, Kheyson S, Lu D, Oparin Y, Kennedy SA, Romerosa B, Arora N, Kwon HY, Jackson K, Prasad M, Jayasekera D, Li A, Guarna G, Natalwalla S, Couban RJ, Reid S, Khan JS, McGillion M, Busse JW. Prevalence and intensity of persistent post-surgical pain following breast cancer surgery: a systematic review and meta-analysis of observational studies. Br J Anaesth. 2020 Sep;125(3):346-357. doi: 10.1016/j.bja.2020.04.088. Epub 2020 Jun 28. PMID 32611524
- [Background] Chen R, Su S, Shu H. Efficacy and safety of rhomboid intercostal block for analgesia in breast surgery and thoracoscopic surgery: a meta-analysis. BMC Anesthesiol. 2022 Mar 16;22(1):71. doi: 10.1186/s12871-022-01599-4. PMID 35296252
- [Background] Elsharkawy H, Saifullah T, Kolli S, Drake R. Rhomboid intercostal block. Anaesthesia. 2016 Jul;71(7):856-7. doi: 10.1111/anae.13498. No abstract available. PMID 27291611

DOCUMENTS (1):
  • Informed Consent Form (2024-12-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT06756048/ICF_000.pdf